CLINICAL TRIAL: NCT06118931
Title: The Impact of Time-restricted Eating, Window Timing, Type 2 Diabetes Status and Sex on Glycemic Control
Brief Title: Time-restricted Eating, Window Timing, Type 2 Diabetes Status and Sex on Glycemic Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Diabetes Canada (Other); Wharton Medical Clinic (Unknown)
Responsible Party: Principal Investigator, Amy Kirkham, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 44122
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Prediabetic State; Hyperglycemia
Keywords: Time-restricted eating; Type 2 Diabetes; Obesity; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Prediabetic State; Hyperglycemia; Intermittent Fasting | interventions — Trehalase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early (7:00-16:00h) TRE (Experimental): Participants will be asked to eat ad libitum between the hours of 7:00 - 16:00 each day for seven days, and then only drink water or other no calorie beverages for the rest of the day. On the 8th day, they will consume one meal replacement beverage at 7:00 and be instructed to not consume anything else for two hours. After the two hours they will be instructed to return to their normal baseline eating habits.
  Interventions: Behavioral: Early (7:00 - 16:00) TRE
- Mid (9:30-18:30h) TRE (Experimental): Participants will be asked to eat ad libitum between the hours of 9:30 - 18:30 each day for seven days, and then only drink water or other no calorie beverages for the rest of the day. On the 8th day, they will consume one meal replacement beverage at 9:30 and be instructed to not consume anything else for two hours. After the two hours they will be instructed to return to their normal baseline eating habits.
  Interventions: Behavioral: Mid (9:30 - 18:30) TRE
- Late (12:00-21:00h) TRE (Experimental): Participants will be asked to eat ad libitum between the hours of 12:00 - 21:00 each day for seven days, and then only drink water or other no calorie beverages for the rest of the day. On the 8th day, they will consume one meal replacement beverage at 12:00 and be instructed to not consume anything else for two hours. After the two hours they will be instructed to return to their normal baseline eating habits.
  Interventions: Behavioral: Late (12:00 - 21:00) TRE
- Control (No Intervention): During the first week of the study, participants will be asked to eat as they normally do, and to not make any changes regarding when they are stopping or starting eating.

INTERVENTIONS:
Behavioral: Early (7:00 - 16:00) TRE — A standardized TRE Protocol where participants eat ad libitum between the hours of 7:00 to 16:00 for 7 days. On the 8th day, they will consume a meal replacement beverage at 7:00, and not consume anything else for two hours.
  Arms: Early (7:00-16:00h) TRE
Behavioral: Mid (9:30 - 18:30) TRE — A standardized TRE Protocol where participants eat ad libitum between the hours of 9:30 to 18:30 for 7 days. On the 8th day, they will consume a meal replacement beverage at 9:30, and not consume anything else for two hours.
  Arms: Mid (9:30-18:30h) TRE
Behavioral: Late (12:00 - 21:00) TRE — A standardized TRE Protocol where participants eat ad libitum between the hours of 12:00 to 21:00 for 7 days. On the 8th day, they will consume a meal replacement beverage at 12:00, and not consume anything else for two hours.
  Arms: Late (12:00-21:00h) TRE

SUMMARY:
This study will evaluate the effectiveness of time-restricted eating (TRE), which is a form of intermittent fasting. When performing TRE, individuals consume all of their calories within a specific time window and then only consume water or other no calorie drinks the rest of the day. TRE is performed each day. There is no restriction on the quality or amount of food that people can consume during their eating window (ad libitum eating) with TRE, which can last anywhere from 4 to 12 hours. We are comparing three different 9-hour eating windows to determine whether the start and stop time of the eating window impact blood sugar control in individuals with obesity who also have or are at risk for type 2 diabetes. We also aim to determine if there are differences in the effects of the timing of eating window between males and females.

DETAILED DESCRIPTION:
The overarching aim of this study is to evaluate the interactions between TRE window timing, type 2 diabetes status, and sex among individuals with obesity. The first objective is to compare the effects of three 9-h TRE window times (early: 7:00-16:00 h, mid: 9:30-18:30 h, delayed: 12:00-21:00 h) on real-time, free-living glycemic control. The second objective is to determine if type 2 diabetes status (type 2 diabetes versus prediabetes or moderate+ risk for type 2 diabetes aka at risk for type 2 diabetes) modifies the effect of eating window timing on glycemic control outcomes. The exploratory objectives include: 1) determine whether sex modifies TRE adherence or the effect of TRE on metabolic changes relative to control; and 2) to compare changes in dietary intake, body weight, and blood pressure within and between early, mid, and delayed TRE. We have the following hypotheses related to these objectives:

1. The early TRE window will result in the most favourable glycemic control outcomes but also the lowest participant acceptability followed by mid and delayed TRE.
2. There will be larger differences in glycemic control outcomes between the TRE window timings among those with type 2 diabetes compared to those at risk for type 2 diabetes.
3. TRE adherence and changes in glycemic control, and weight loss with all TRE window times (relative to control) will be higher in men vs women.
4. Energy, carbohydrate, and sugar intake, body weight, and blood pressure will decrease during TRE, but with no differences by window timing.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Body mass index >30 kg/m2 and <50 kg/m2
* Have access to an Apple or Android cellphone with Bluetooth.
* Have type 2 diabetes or be at risk for type 2 diabetes (defined as high (33+) Canadian Diabetes Risk Score)

Exclusion Criteria:

* Individuals with type 2 diabetes will be excluded if: (1) currently on >3 monotherapies for diabetes, (2) have had diabetes therapy dosage changes <3 months, (3) self-reported hemoglobin A1c >9.0%, (4) taking exogenous insulin, or (5) taking sulfonylureas
* The following exclusion criteria applies to all potential participants:

  1. History of or referral for bariatric surgery
  2. Weight loss >5% in the last 3 months
  3. Taking antiobesity (weight loss) medications
  4. Body weight >340lbs
  5. Diagnosed cognitive disorder that precludes them from giving consent
  6. Inability or unwillingness to change their eating window to follow those prescribed in the study
  7. Currently eating during <12 hour period on 5 or more days/week
  8. Physician-diagnosed eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Average 24-hour glucose total area under the curve (AUC) over 7 days | 7 days
  Assessed for 7 continuous days using a continuous glucose monitor.

SECONDARY OUTCOMES:
Average 24-hour glucose over 7 days | 7 days
  Assessed for 7 continuous days using a continuous glucose monitor.
Average daily nocturnal glucose over 7 evenings | 7 days
  Assessed for 7 continuous evenings based on the sleep period identified by the Fitbit tracker using a continuous glucose monitor.
Average daily time spent in hyperglycemia over 7 days | 7 days
  The average number of hours with glucose >10 mmol/L over 7 continuous days assessed with a continuous glucose monitor.
Postprandial glucose | 2 hours
  Assessed on the morning after the 7th day of each TRE protocol. Participants will consume a standardized breakfast at a specified time, and glucose will be evaluated via continuous glucose monitor from the time they start consuming the breakfast for 2 hours.
Glycemic viability | 7 days
  The average of each standard metrics of glycemic viability (standard deviation, coefficient of variation, mean amplitude of glycemic exercise, and continuous overall net glycemic action) will be calculated over 7 continuous days from continuous glucose monitors.
Patient acceptability | 7 days
  Patient acceptability will be assessed based on researcher-developed questions related to their experience with each TRE protocol.
TRE fasting duration adherence | 7 days
  Participants will receive twice daily text messages asking what time they started and stopped eating that day, which will be used to calculate the length of the fast each day. Adherence will be calculated as the % of days where the participant fasted for 15h or longer.
TRE fasting window adherence | 7 days
  The proportion of days where participants began and ended their meal within 15 min or 30 min of their prescribed time.

OTHER OUTCOMES:
Dietary intake | 7 days
  Participants will complete the ASA-24 at baseline, and during each of the intervention periods to assess changes in macro and micronutrient composition of their diet.
Weight change | 7 days
  Participants will be asked to weigh themselves first thing in the morning, with minimal and no clothing on, after they have emptied their bowels once during the baseline period and on the last day of each of the intervention period.
Blood pressure change | 7 days
  Participants will be asked to measure their blood pressure once during the baseline period, and on the last day of each intervention period.
Physical Activity | 7 days
  Participants will be asked to wear a Fitbit for the duration of the study. We will average the amount of physical activity over 7 days of wear.
Sleep | 7 days
  Participants will be asked to wear a Fitbit for the duration of the study. We will average the amount of sleep over 7 days of wear.
Safety and Adverse Events | 7 days
  Participants will be given access to a questionnaire to report any symptoms throughout the intervention. We will compare the proportion of individuals who report these symptoms within each time period.

CONTACTS AND LOCATIONS:
Overall Officials: Amy A. Kirkham, PhD, Principal Investigator — University of Toronto
Locations (1):
- Remote Ontario-wide, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No